CLINICAL TRIAL: NCT07241338
Title: Sacubitril/Allisartan Versus Amlodipine for Hypertensive Patients With Overweight or Obesity: A Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: Sacubitril/Allisartan for Hypertensive Patients With Overweight or Obesity
Acronym: SHOT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jing Liu (Other)
Responsible Party: Sponsor-Investigator, Jing Liu, Director of the Department of Hypertension, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025PHB414
Record Dates: First submitted 2025-11-13; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: obesity; overweight; hypertension; sacubitril/Allisartan
MeSH Terms: conditions — Hypertension; Obesity; Overweight | interventions — sacubitril; Amlodipine; Calcium Channel Blockers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/Allisartan (Experimental)
  Interventions: Drug: sacubitril/allisartan
- Amlodipine (Active Comparator)
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: sacubitril/allisartan — Oral administration of sacubitril/allisartan 240mg once daily for 4 consecutive weeks. If blood pressure reaches the target, the original regimen is continued; otherwise, the dose of sacubitril/valsartan is increased to 480mg once daily for another 4 weeks of treatment
  Other Names: angiotensin receptor neprilysin inhibitor; ARNI
  Arms: Sacubitril/Allisartan
Drug: Amlodipine — Amlodipine group: Oral administration of amlodipine 5mg once daily for 4 consecutive weeks. If blood pressure reaches the target, the original regimen is continued; otherwise, the dose of amlodipine is increased to 10mg once daily for another 4 weeks of treatment
  Other Names: calcium channel blocker; CCB
  Arms: Amlodipine

SUMMARY:
To compare the efficacy and safety of sacubitril/Allisartan versus amlodipine in the antihypertensive treatment of overweight/obese patients with primary hypertension

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled, open-label trial conducted in overweight/obese patients with primary mild-to-moderate hypertension, aiming to compare the efficacy and safety of sacubitril/Allisartan versus amlodipine treatment.

The study consists of two phases: a washout period (maximum 2 weeks, for patients currently receiving antihypertensive medication) and a treatment period (8 weeks). Patients already on antihypertensive therapy must complete a 2-week washout period (i.e., discontinue antihypertensive treatment), while those with no prior history of antihypertensive medication use are exempt from the washout.

All patients undergo eligibility assessment against inclusion and exclusion criteria before randomization. Eligible patients are randomly assigned in a 1:1 ratio to sacubitril/Allisartan group or Amlodipine group. In sacubitril/Allisartan group, oral administration of sacubitril/Allisartan 240mg once daily for 4 consecutive weeks. If blood pressure reaches the target, the original regimen is continued; otherwise, the dose of sacubitril/Allisartan is increased to 480mg once daily for another 4 weeks of treatment. In Amlodipine group, oral administration of amlodipine 5mg once daily for 4 consecutive weeks. If blood pressure reaches the target, the original regimen is continued; otherwise, the dose of amlodipine is increased to 10mg once daily for another 4 weeks of treatment.

The total treatment period is 8 weeks of oral medication. Patients will attend study visits on the day before treatment initiation (Day 0), at the end of Week 4, and at the end of Week 8 of the treatment period for efficacy and safety assessments, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years inclusive, regardless of gender;
2. Body Mass Index (BMI) ≥ 24 kg/m²;
3. Diagnosed with essential hypertension, either untreated or currently receiving antihypertensive medication;
4. For patients who have not received antihypertensive medication in the past 3 months, the msSBP at the screening visit must be ≥ 150 mmHg and < 180 mmHg;
5. For patients currently receiving antihypertensive medication, the msSBP at the screening visit must be ≥ 140 mmHg and < 180 mmHg; and at the visit after the washout period, the msSBP must be ≥ 150 mmHg and < 180 mmHg.

Exclusion Criteria:

1. Severe hypertension (msSBP ≥ 180 mmHg and/or msDBP ≥ 110 mmHg); malignant hypertension, etc.;
2. History of or diagnostic evidence for obstructive sleep apnea (OSA);
3. History of angioedema;
4. History of or diagnostic evidence for secondary hypertension;
5. Hypertension complicated with the following conditions: acute coronary syndrome, myocardial infarction, percutaneous coronary intervention, or stroke occurring within 12 months; New York Heart Association (NYHA) Class II-IV heart failure, large aortic aneurysm or aortic dissection, atrioventricular block of degree II or higher, sick sinus syndrome, bradycardia (heart rate < 50 beats per minute) or other arrhythmias requiring antiarrhythmic drugs, as well as severe diseases such as epilepsy and syncope;
6. Clinically significant abnormalities in laboratory tests (serum potassium > 5.5 mmol/L or < 3.5 mmol/L; serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2.5 × upper limit of normal (ULN); serum creatinine > 1.5 × ULN);
7. Type 1 diabetes mellitus and type 2 diabetes mellitus with poor glycemic control (glycated hemoglobin (HbA1c) > 8.0%);
8. Patients currently using drugs with weight-loss effects such as glucagon-like peptide-1 (GLP-1) and sodium-glucose cotransporter 2 (SGLT-2) inhibitors;
9. Patients undergoing hemodialysis or strict salt-restriction therapy;
10. Known or suspected allergy to sacubitril/allisartan, sacubitril/valsartan sodium, amlodipine, or related drugs;
11. Patients deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The change in the mean sitting systolic blood pressure (msSBP) from baseline to week 8, assessed for sacubitril/allisartan as compared to amlodipine | From the start of randomization to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
The change in the mean sitting diastolic blood pressure (msSBP) from baseline to week 8, assessed for sacubitril/allisartan as compared to amlodipine | From the start of randomization to the end of treatment at 8 weeks
The BP control rate of sacubitril/allisartan compared to amlodipine | From the start of randomization to the end of treatment at 4 weeks and 8 weeks
  BP control was defined as msSBP/msDBP < 140/90mmHg
The BP response rate of sacubitril/allisartan compared to amlodipine | From the start of randomization to the end of treatment at 8 weeks
  The percentage of patients who had a successful response after treatment for msSBP (<140 mmHg or a reduction by ≥20 mmHg from baseline) and msDBP (<90 mmHg or a reduction by ≥10 mmHg from baseline)
Changes in 24-hour mean ambulatory systolic and diastolic blood pressures of sacubitril/allisartan compared to amlodipine | From the start of randomization to the end of treatment at 8 weeks
Changes in daytime and night-time mean ambulatory blood pressures of sacubitril/allisartan compared to amlodipine | From the start of randomization to the end of treatment at 8 weeks
Changes in circadian rhythm of blood pressure between sacubitril/allisartan compared to amlodipine | From the start of randomization to the end of treatment at 8 weeks
Safety assessments between sacubitril/allisartan compared to amlodipine | From the start of randomization to the end of treatment at 8 weeks
  Number of participants with adverse events (AEs), serious AEs (SAE), adverse drug reactions (ADR), with abnormal vital signs, abnormal physical exam findings, abnormal laboratory tests results

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No